CLINICAL TRIAL: NCT04682535
Title: Daily Study of Caregiving Relationships and Health
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: HSC20200421H
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Caregiver Burnout; Dementia; Dementia of Alzheimer Type; Relations, Family; Social Stress; Relation, Interpersonal; Loneliness
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples from a subsample of n=11 caregivers retained, including 4 samples/day for 5 days per caregiver.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Spousal/partner family caregivers to persons living with dementia. Participants will complete 14-days of surveys about their relationships, social interactions, as well as health and health behaviors. A subsample of n=15 may volunteer to provide diurnal saliva samples.
  Interventions: Other: Social relationships

INTERVENTIONS:
Other: Social relationships — Exposure to social interactions with spouse, friends, and family. Perceived loneliness, emotional strain, and emotional support.

SUMMARY:
The purpose of the Daily Study of Caregiving Relationships and Health is to learn how caregiving relationships and social connectedness are associated with dementia caregivers' health, health behaviors, and diurnal patterns of salivary cortisol.

This is a pilot study wherein the purpose is to test the feasibility and acceptability of study protocols.

DETAILED DESCRIPTION:
The purpose of the Daily Study of Caregiving Relationships and Health is to learn how caregiving relationships and social connectedness are associated with dementia caregivers' health, health behaviors, and diurnal patterns of salivary cortisol. Investigators are asking caregivers to complete 14-days of surveys which ask about their relationships and health behaviors, in addition to 2 longer surveys (baseline and 3-month follow up). Investigators hypothesize that on days when caregivers receive more emotional support, they will report better health behaviors (e.g., improved sleep quality). On days when caregivers experience greater 1) strain and 2) loneliness, they will report poorer health behaviors. Information about which aspects of social relationships and social connectedness most affect health will be used to inform interventions programs.

ELIGIBILITY:
Inclusion Criteria:

* Spouse or partner to an individual living with ADRD who has received a diagnosis from a physician
* Aged 18 years or older Provides assistance with at least one instrumental activities of daily living or activities of daily living
* Not paid to provide care
* Cares for someone with a global deterioration score of 1 to 5 (early to mid-stage dementia)
* Has reliable access to email and text messaging, and smart phone device
* Live within 40 miles of UT Health San Antonio (if completing saliva collection protocol)

Exclusion Criteria:

* Inability to read and speak English or Spanish
* Vision or hearing impairment affecting ability to complete study protocols (e.g., blindness)

Additional exclusion Criteria if completing saliva collection protocol:

* Experiencing a major health event within the previous 6 months (e.g., stroke, myocardial infarction, in-patient surgery, cancer besides skin cancer)
* Symptoms of infectious disease within the previous 14-days (e.g., COVID-19, oral infection)
* Diagnosis of major depressive disorder
* HPA axis endocrine disorder (e.g., Cushings or Addison's disease)
* Use of corticosteroid medication
* Pregnancy
* Participation in overnight shift work

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Spousal family caregivers to persons diagnosed with dementia (any type)
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Frequency of daily health symptoms | 2 weeks
  Frequency of adverse health symptoms experienced by participant (e.g., fatigue; 0 to 21)
Perceived sleep quality | 2 weeks
  Perceived sleep quality the night prior (1 to 5)
Physical activity | 2 weeks
  Participation in at least 30 minutes of moderate to vigorous physical activity (binary)
Consumption of alcoholic beverages | 2 weeks
  Consumption of 1 or more alcoholic beverages (binary)
Potential binge eating behaviors | 2 weeks
  Frequency of binge eating behaviors, including consuming unusually large amount of food, feeling out of control, and unplanned and repetitive eating (0 to 33)

SECONDARY OUTCOMES:
Total salivary cortisol | 2 weeks
  Area under the curve score to approximate total cortisol output during the day (μg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD used for publication will be available by contacting (i.e., emailing) the PI. Supporting materials available upon request and at PI's discretion.
Time Frame: IPD available following publication of peer-reviewed manuscripts and made available to peer-reviewers upon request